CLINICAL TRIAL: NCT07229443
Title: Evaluation of a Colorectal Cancer Education Training Program
Brief Title: CoGENES Randomized Controlled Trial (RCT)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19PS-24-7; NCI-2025-02815 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19PS-24-7 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH); U2CCA252971-01 (NIH)
Record Dates: First submitted 2025-09-16; First posted 2025-11-17 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Health Promotion; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (usual care) (Active Comparator): Participants receive a packet of existing information materials about colorectal cancer prevention, screening, and genetic testing to review at their own pace over 6-10 weeks. Participants may optionally receive a CoGENES training session within 2 weeks post-intervention.
  Interventions: Other: Best Practice; Other: Survey Administration
- Group 2 (CoGENES) (Experimental): Participants receive a CoGENES training session over 45-60 minutes.
  Interventions: Other: Health Promotion and Education; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive a packet of existing information materials about colorectal cancer prevention, screening, and genetic testing
  Other Names: standard of care; standard therapy
  Arms: Group 1 (usual care)
Other: Health Promotion and Education — Receive CoGENES training
  Arms: Group 2 (CoGENES)
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates the effectiveness of trained community engagement specialists for improving communication on colorectal cancer (CRC) prevention and genetic testing among Hispanic/Latino/a/x (H/L) communities. CRC is the second and third leading cause of cancer deaths among United States (US) H/L men and women respectively. Knowledge of inherited germline mutations (changes in a gene that occurs in a sperm or egg cell) is critical for understanding cause of disease and can impact patient treatment options and outcomes. Educational programs and participant engagement approaches focused on H/L individuals considering Latino cultural values, literacy, numeracy, barriers faced, cultural beliefs and attitudes, as well as language of participants are much needed to address these observed disparities. The Community Genetic Navigation Specialists (CoGENES) Program focuses on increasing knowledge, and preparing the CoGENES trainees to help respond to questions, fears, and concerns regarding genetic testing, counseling, biospecimen (sample of urine, blood, or tissue cells) donation and participation in clinical trials to H/L community members, patients and their families. CoGENES may improve communication on colorectal cancer prevention and genetic testing which can help reduce cancer disparities among H/L communities.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To develop a local workforce of trained community engagement specialists to act as liaison agents to improve communication on genetic research, clinical genetic testing, and counseling to Hispanic/Latino/a/x (H/L) individuals.

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP 1: Participants receive a packet of existing information materials about colorectal cancer prevention, screening, and genetic testing to review at their own pace over 6-10 weeks. Participants may optionally receive a CoGENES training session within 2 weeks post-intervention.

GROUP 2: Participants receive a CoGENES training session over 45-60 minutes.

After completion of study intervention, participants are followed up at 8 weeks, 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older
* Ability to understand and the willingness to sign a written informed consent
* Self-reported H/L ethnicity, of any race
* Ability to read, write, and speak Spanish or English
* Resides in Los Angeles County

Exclusion Criteria:

* Anyone younger than 18 years of age
* Any person with major cognitive deficit or psychiatric impairment
* Any person unable to read and write Spanish or English
* Resides outside of Los Angeles County
* Any person who considers themselves a community health educator or "promotor/a de salud" and/or has taken in the past three years training on colorectal cancer and/or cancer genetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Change in knowledge about colorectal cancer prevention | Baseline to 12 months
  We will use the WCRF/AICR score, which is a standardized scoring system, typically ranging from 0 to 7 points, that measures an individual's adherence to the World Cancer Research Fund (WCRF) and American Institute for Cancer Research (AICR) recommendations for cancer prevention. A higher score indicates greater compliance with lifestyle factors like maintaining a healthy weight, engaging in physical activity, eating a diet rich in plant-based foods, and limiting alcohol, fast food, and sugary drinks. We will compare pre- and post-intervention to assess knowledge.
Change in knowledge about genetic testing | Baseline to 12 months
  Will use the Genetic Literacy and Comprehension (GLAC) measure to assess participant knowledge with eight commonly used genetic terms and concepts (genetic, chromosome, susceptibility, mutation, variation, abnormality, heredity, and sporadic) using a 7-point scale of 1 "Strongly Disagree" to 7 "Strongly Agree". We will compare pre- and post- surveys to assess knowledge.
Change in knowledge about tumor testing | Baseline to 12 months
  Will assess participants knowledge about tumor testing as determined by scores obtained from validated surveys. Will compare pre- and post- surveys to assess knowledge. Higher scores mean better knowledge.
Change in knowledge about genetic counseling | Baseline to 12 months
  There are 14 items in the questionnaire of Cancer Genetic Knowledge Scale. The total score ranges between 14 and 70. Higher scores indicate more/better knowledge. The questionnaire will be administered at pre- and post-genetic education.
Changes in dietary and lifestyle patterns | Baseline to 12 months
  Measured by scores obtained from surveys developed for this study. Will compare pre- and post- surveys to evaluate changes. Higher scores mean positive changes.
Intention to pursue colorectal cancer screening | Up to 12 months
  Will be assessed using one question with a 5-point response option (1 = Very Unlikely, 2 = Somewhat Unlikely, 3 = Neutral, 4 = Somewhat Likely, 5 = Very Likely).
Intention to inquire about cancer history among family members | Up to 12 months
  Will be assessed using one question with a 5-point response option (1 = Very Unlikely, 2 = Somewhat Unlikely, 3 = Neutral, 4 = Somewhat Likely, 5 = Very Likely).
Intention to ask healthcare provider about genetic testing and counseling | Up to 12 months
  Will be assessed using one question with a 5-point response option (1 = Very Unlikely, 2 = Somewhat Unlikely, 3 = Neutral, 4 = Somewhat Likely, 5 = Very Likely).

CONTACTS AND LOCATIONS:
Overall Officials: Mariana C Stern, PhD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States